CLINICAL TRIAL: NCT04534751
Title: Prospective, Multi-center, Randomized, Parallel-control, Superiority Study Comparing Administration of Clotting Factor Concentrates With a Standard Massive Hemorrhage Protocol in Severely Bleeding Trauma Patients.
Brief Title: Factor In the Initial Resuscitation of Severe Trauma 2 Patients
Acronym: FiiRST-2
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Recruiting
Sponsor: University Health Network, Toronto (Other)
Collaborators: Sunnybrook Health Sciences Centre (Other); Octapharma (Industry); Canadian Institutes of Health Research (CIHR) (Other Government); Canadian Institute for Military and Veteran Health Research Defense Research & Development Canada (Unknown)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: 20-5828; 2031 (CTO ID) (Other: Sunnybrook Health Sciences Centre)
Record Dates: First submitted 2020-08-27; First posted 2020-09-01 (Actual); Last update posted 2022-12-05 (Actual); Status verified 2022-12

CONDITIONS: Traumatic Hemorrhage; Coagulopathy; Massive Hemorrhage
Keywords: Trauma; Injury; Acute trauma coagulopathy; Traumatic bleeding; Clotting factors; Fibrinogen; Fibrinogen concentrate; Prothrombin complex concentrate; Massive Hemorrhage Protocol; Frozen Plasma
MeSH Terms: conditions — Hemostatic Disorders; Wounds and Injuries; Hemophilia B | interventions — Fibrinogen; prothrombin complex concentrates

STUDY DESIGN:
Intervention Model Description: Prospective, multi-center, randomized, parallel-control, superiority study comparing administration of clotting factor concentrates with a standard massive hemorrhage protocol in severely bleeding trauma patients.
Who Masked: Participant, Investigator, Outcomes Assessor
Masking Description: Given blood products in each randomized arm have different physical differences, it is not possible to blind the treating health care providers to group assignment.
  Clinicians not involved in the acute resuscitation period (MHP activations usually last under 4 hours) and outcome assessors will remain blinded by using a generic product label in the patient chart and/or the electronic product name (i.e., FiiRST-2 MHP pack 1 and pack 2, rather than specifying type of product used). The first pack will be sealed, and the treating health care providers will be instructed to refrain from opening the first pack until the decision is made to transfuse clotting factor replacement.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Intervention Group- Clotting Factor Concentrates (Experimental): Fibryga + Octaplex (Fibrinogen + PCC)
  Fibrinogen Concentrate 4g (Fibryga) + Prothrombin Complex Concentrate 2000 IU (Octaplex) in the first and second massive hemorrhage protocol (MHP) packs.
  Interventions: Biological: Fibrinogen + PCC
- Control Group: Standard FP transfusion (Active Comparator): Frozen Plasma (FP)
  Interventions: Biological: Frozen Plasma

INTERVENTIONS:
Biological: Fibrinogen + PCC — Patients randomized to the intervention group will receive 4g of Fibryga and 2000 IU Octaplex will be released as part of the first and second MHP packs, if requested.
  If a third MHP pack is required, and thereafter, FC will be administered if the fibrinogen level drops below 1.5-2.0 g/L at the discretion of the clinical team or based on conventional laboratory test results or viscoelastic methods.
  Patients in both groups will otherwise receive identical MHP treatment packs (4 units of red blood cells [RBC] in pack 1 and 4 units of RBC and 1 pool of platelets in pack 2 (equivalent to 4 units).
  Other Names: Fibryga + Octaplex
  Arms: Intervention Group- Clotting Factor Concentrates
Biological: Frozen Plasma — 4U FP will be released as part of the first and second MHP packs.
  Patients in both groups will otherwise receive identical MHP treatment packs (4 units of red blood cells [RBC] in pack 1 and 4 units of RBC and 1 pool of platelets in pack 2 (equivalent to 4 units).
  Patients randomized to the control group may receive FC if the fibrinogen level drops below 1.5-2.0 g/L at the discretion of the clinical team or based on conventional laboratory test results or viscoelastic methods. FC dosing in MHP packs 3 and above will be site-specific and at the discretion of the treating clinician.
  Arms: Control Group: Standard FP transfusion

SUMMARY:
Injury is the leading cause of death for people between the ages of 1-44. This is especially true in trauma patients who have bleeding complications. Acute trauma coagulopathy (ATC) is associated with high transfusion requirements, longer ICU stays, and a greater incidence of multi-organ dysfunction. The cause of coagulopathy is multi-factorial.

One major driver is acquired fibrinogen deficiency (hypofibrinogenemia). Fibrinogen is critical in clot formation and enhances platelet aggregation. Due to the body's limited reserve, it is the first clotting factor to fall to critical levels during life-threatening bleeding. This can impair coagulation and increases bleeding complications. There are two primary options available for fibrinogen supplementation:

* Cryoprecipitate- North American standard
* Fibrinogen Concentrate (FC)- European standard

Consumption of coagulation factors, including fibrinogen, is another important component of ATC. To replenish these depleted coagulation factors and improve thrombin generation, two therapies are available:

* Frozen Plasma (FP)- North American standard
* Prothrombin Complex Concentrate (PCC)- European standard

Strategies for hemorrhage and coagulopathy treatment have changed significantly over the last decade. Prompt hemorrhage control, along with targeted coagulation factor replacement, are emerging as key components of trauma care. Currently, the initiation of a massive hemorrhage protocol (MHP) results in red blood cells (RBCs) and FP transfusions in a 1:1 or 2:1 ratio. Clotting factors are replaced via FP administration. Fibrinogen supplementation is administration after lab verification or at the clinician's discretion. MHP continues until the rate of hemorrhage is under control.

FC and PCC have several important advantages over cryoprecipitate and FP but there is a scarcity of data regarding their efficacy and safety of their use in hemorrhaging trauma patients. The FiiRST-2 study aims to understand if early use of FC and PCC in trauma patients at risk of massive hemorrhage will lead to superior patient outcomes. This trial will also provide safety data on early administration of FC and PCC as a first-line hemostatic therapy in trauma care, and its impact on hemostatic and other clinical endpoints.

DETAILED DESCRIPTION:
Study Design and Duration FiiRST-2 is a multicenter, randomized, parallel-control, superiority trial, utilizing a conventional two-armed, two-stage design, with an adaptive interim analysis, performed at Level 1 Trauma Centers in Canada. The study is designed to examine the effect of replacing fibrinogen and clotting factors via FC and PCC following activation of the massive hemorrhage protocol (MHP) on the number of ABP units transfused in trauma patients with severe hemorrhage versus the current standard of care (ratio-based plasma resuscitation).

Test Products, Dose, and Mode of Administration:

Patients will be randomized if the MHP is activated according to the MHP activation criteria at each study site. Once eligibility is confirmed, the blood bank medical laboratory technologist will randomize the patient to one of two groups: the intervention group or the control group.

* Intervention group: 4 g Fibryga and 2000 IU Octaplex will be released as part of the first and second MHP packs.
* Control group: 4 U FP will be released as part of the first and second MHP packs.
* Concomitant therapy: In both groups, 4 U RBC will be included as part of the first and second MHP packs, and 1 dose of platelets (4 U of pooled random donor or single donor apheresis) will also be included as part of the second MHP pack. Both RBCs and platelets will be administered according to the clinical situation and/or lab results as per the discretion of the clinical team. The second MHP pack will be released at the request of the clinical team, but clinicians will be instructed to administer all of the investigational product (Fibryga/Octaplex or FP) in the first pack before moving onto the second pack. Similarly, if the second pack is opened, clinicians will be instructed to administer all of the investigational products contained within, before moving to the third pack. Not administering all of the investigational products in the first pack, once started, will be a protocol deviation.

Administration of all non-investigational products will be at the discretion of the clinical team according to the hemodynamic status of the patient and/or laboratory results (standard and/or point-of-care as per institutional practice). While platelets will be routinely included in the second pack, clinicians can request platelets outside of the packs (e.g., for patients on antiplatelet therapy or with marked thrombocytopenia). In the control group, FC may be administered if hypofibrinogenemia (fibrinogen level below 1.5-2.0 g/L or FIBTEM A10 below 8-12 mm) is identified as part of routine testing, at the discretion of the clinical team. Patients in the intervention group can receive additional FC if hypofibrinogenemia (as per above criteria) is identified after the full dose (4g) in the first pack is administered (if the second pack is not opened). If the second pack is opened, additional doses of FC will be permitted after the full dose (4g) in the second pack is administered..

Patients in the control group will not be permitted to receive PCC during the study. Patients in the intervention group may receive FP in the third and subsequent MHP packs. If a third MHP pack is required, and thereafter, MHP packs will contain ABPs (RBCs, platelets and plasma) according to guidelines at each participating site or revert to laboratory-guided transfusion as per the local guidelines once bleeding is controlled. The MHP should be terminated once bleeding is controlled and the MHP criteria are no longer met. Termination of the MHP may occur at any time based on the discretion of the clinical team.

The maximum time frame for administration of the second MHP pack (if required) for both groups is 24 hours from arrival to the trauma bay/ED or termination of the MHP (whichever comes first).

We anticipate for the trial to begin in June 2020 and be completed over a 3 year period.

Sample Size The study will enroll up to 350 trauma patients with approximately 175 assigned to each of the two treatment groups.

Due to the inherent variability in the primary endpoint and a yet substantial uncertainty about the effect size, an adaptive design approach will be used. For this, a planned interim analysis will be performed after 120 patients have completed the study at up to four hospital sites. Primary aim of this interim analysis is to calculate the p-value and conditional power of the test statistic and perform a sample size re-assessment. This will be done in an unblinded interim analysis performed by an independent statistician who will report the results only to the independent data safety monitoring committee (IDSMC) which will make recommendations to the sponsor without revealing the treatment groups. Hence, the final number of enrolled patients will depend on the sample size re-calculation.

ELIGIBILITY:
Inclusion Criteria:

Severely injured adult trauma patients who meet all following criteria:

1. Estimated age greater than 16 years old
2. Severely injured (penetrating or blunt) trauma patients
3. Triggered MHP within first hour of hospital arrival at the trauma bay/ED

Exclusion Criteria:

Patients who meet any of the following criteria are not eligible for the study:

1. Have received more than 2 U RBCs during the pre-hospital phase of care
2. Have received more than 2 U RBCs in the trauma bay/ED before activation of the MHP
3. Have an elapsed time from injury of more than 3 hours
4. Have a penetrating traumatic brain injury with Glasgow Coma Scale (GCS) of 3
5. Are suspected or known to be on anticoagulants in the last 7 days
6. Have known congenital or acquired bleeding disorders
7. Have a known pregnancy
8. Refuse blood transfusion due to religion or other reasons
9. Previous history of heparin induced thrombocytopenia (HIT)

Min Age: 16 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2021-04-01 (Actual); Primary Completion 2023-12-31 (Estimated); Study Completion 2024-01-30 (Estimated)

PRIMARY OUTCOMES:
Composite of total number of Allogeneic Blood Products (ABPs) | within 24 hours
  The primary endpoint is to demonstrate superiority with respect to the composite number of all ABP units (RBCs, FP and platelets) transfused

SECONDARY OUTCOMES:
Total number of RBC units | Transfused within the 24 hours
  RBC - Red Blood Cells
Incidence of thromboembolic events | up to 28 days
  Defined by evidence of any of the following:
  * Deep vein thrombosis (DVT)
  * Pulmonary embolism (PE)
  * Myocardial infarction (MI)
  * Ischemic stroke o. Arterial or venous thrombosis at other sites
Ventilator-free days | From arrival to day 28
  defined as the number of days up to Day 28 following arrival at the trauma bay/ED on which a patient breathed without assistance (if period of unassisted breathing lasted at least 48 consecutive hours). Patients who die during study follow-up or require 28 or more days of mechanical ventilation will be assigned zero ventilator-free days

CONTACTS AND LOCATIONS:
Overall Officials: Luis T Da Luz, MD, Principal Investigator — Sunnybrook Health Sciences Centre
Locations (6):
- Canada (6):
  - Vancouver General Hospital, Vancouver, British Columbia
  - Hamilton Health Sciences and McMaster University, Hamitlon, Ontario
  - Kingston Health Sciences Centre, Kingston, Ontario
  - Victoria Hospital, London, Ontario
  - Sunnybrook Health Sciences Centre, Toronto, Ontario
  - St. Michael's Hospital, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No
No current plan to make IPD available to other researchers.

REFERENCES:
- [Derived] da Luz LT, Karkouti K, Carroll J, Grewal D, Jones M, Altmann J, Lin Y, Gupta A, Nathens AB, Kron A, Notario L, Beckett A, Petrosoniak A, Pavenski K, Vogt K, Ball IM, Parry NG, Engels PT, Zeller MP, Arnold DM, Belley-Cote E, Evans C, Leitch J, Shih A, Dawe PJ, Gooch R, Callum J. Factors in the Initial Resuscitation of Patients With Severe Trauma: The FiiRST-2 Randomized Clinical Trial. JAMA Netw Open. 2025 Sep 2;8(9):e2532702. doi: 10.1001/jamanetworkopen.2025.32702. PMID 40982282
- [Derived] da Luz LT, Callum J, Beckett A, Hucke HP, Carroll J, Grewal D, Schwartz B, Peng H, Engels PT, Parry N, Petrosoniak A, Tien H, Nathens AB, Scales D, Karkouti K. Protocol for a multicentre, randomised, parallel-control, superiority trial comparing administration of clotting factor concentrates with a standard massive haemorrhage protocol in severely bleeding trauma patients: the FiiRST 2 trial (a 2020 EAST multicentre trial). BMJ Open. 2021 Sep 3;11(9):e051003. doi: 10.1136/bmjopen-2021-051003. PMID 34479938